CLINICAL TRIAL: NCT04749121
Title: Impact of Ultraviolet Germicidal Irradiation on the New Silicone Half-Piece Elastometric Respirators (VJR-NMU) Respirator Performances, Structural Integrity and Sterility During COVID -19 Pandemic:
Brief Title: Ultraviolet Germicidal Irradiation on the New Silicone Half-Piece Elastometric Respirators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 059/63
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: COVID-19; Decontamination; Filtering facepiece respirators; UVC
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Before and after intervention in one group
Masking Description: The participants will be tested for fit test before and after UVC determination of the respirators.The other tests were in vitro and based on the survival of bacteria and virus on the masks together with the tensile strength
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fit test (Experimental): All the participants had to pass the initial fit test.After decontamination with UVC irradiation for 60 minutes.The protocol was conducted in accordance with the protocol from the OSHA respiratory protection standard , including the number, type, and duration of the exercise, and the seal checks in accordance with the manufacturer's instructions[15] 60 minutes, fit testing was conducted using qualitative fit test (Bittrex Solution aerosol)
  Interventions: Device: UVC Irradiation; Drug: UVC Irradiation; Device: Fit test; Device: Tensile strength

INTERVENTIONS:
Device: UVC Irradiation — We used the Porcine epidemic diarrhea virus (PEDV) as the indicator virus .An N99 mask was contaminated by spraying or applying with the virus on the exterior and interior surface of each silicone mask. Also, 100 μl of the viral suspension was spotted onto the filter part of N99 masks. Following 20-30 minutes of drying, the silicone masks underwent each of the decontamination procedures which are ultraviolet-C (UV-C) irradiation and 70% alcohol treatment. For UV irradiation, N99 masks were placed in an UV-C incubator ) and were exposed for different times at 1, 10 and 20 minutes, respectively.Untreated control and treated N99 masks were analyzed for viral infectivity in VERO cell cultures. At 48 hours post-infection, cells were examined for evaluation the viral infectivity via observation of cytopathic effect. Results for each treatment express mean ± standard deviations of 3 biological replicates.
Drug: UVC Irradiation — Bacterial and fungal sampling were obtained from the inside and outside surface areas likely to the frequently touched and close contact with the face of hospital personnel. The cultures were then isolated onto the blood agars and Mac Conkey agars, respectively. After incubation, the total number of bacterial and fungal colonies were counted, recorded, and selected different colonies.
Device: Fit test — All the participants had to pass the initial fit test.After decontamination with UVC irradiation for 60 minutes, fit testing was conducted using qualitative fit test (Bittrex Solution aerosol),
Device: Tensile strength — We measured the tensile strength of the strap of the Silicone mask before and after the UVC irradiation to study the strength and reliliency of the strap

SUMMARY:
Since the innovation of our new half- elastometric half-piece respirator, this type of FFR has been used widely in our country. Decontamination methods including ultraviolet C (UVC) germicidal irradiation and 70% alcohol have been implemented to decontaminate the respirator. We than examined inactivation potential for the Porcine epidemic diarrhea virus (PEDV), numerous bacterial strains ,mostly skin-derived after the decontamination process.To enable rigorous integrity after repeated decontamination process, fit test by the Bitrex test ,tensile strength and elongation at break were also evaluated. Our results showed that the UVC at the dose of 3 J/cm2 can eradicate the bacteria at 60 min and virus at 10 min.No fungus was found on the mask surface at the beginning. Good Fit test , tensile strength and elongation at break were still main maintained after multiple cycles of decontamination. No evidence of physical degradation by gross visual inspection was found. 70% alcohol is also an easy and effective way to eradicate microorganisms on the mask.As the current pandemic is expected to continue for months to years, the need to supply adequate reserves of PPE and develop effective reprocessing is crucial. Our studies demonstrated that the novel silicone mask can be safely reprocessed and decontaminated for many cycles by UVC irradiation and help restore the shortage of the important protective devices in the COVID-19 pandemic era.

DETAILED DESCRIPTION:
this study showed that UVC irradiation at the dosage 300 uWatt-sec/cm2 for 1 minute satisfactorily decontaminated the silicone mask as measured by viral culture. The timing to eradicate bacteria was 60 minutes longer due to the tolerability of the bacteria .70% alcohol effectively decontaminate the virus and bacteria deposited on the masks and filters. Good level of fit can be maintained following UVC treatment. The tensile strength of the strap was retained over multiple decontamination cycles using UVC and dry heat upto 60 cycles.Given the efficacy of the disinfection by UVC and 70 % alcohol ,these types of decontamination method could potentially be used for the new type of silicone masks half-piece respirator in the setting of a crisis with inadequate supplies of PPE.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers 18 to 60 years old.

Exclusion Criteria:

* contraindications to fit test, such as asthma, congestive heart failure, anosmia, and ageusia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Fit test | 3 days
  The percent of participants that passed the fit test after UVC decontamination
Colony count of microorganisms | 2 weeks
  Colony count of virus ,bacteria and fungus after UVC and alcohol decontamination
Load of Tensile strength | 2 weeks
  Measure tensile strength and elengation at break after UVC irradiation (Millipascal)

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, Principal Investigator — Bangkok Metropolitan Administration and Vajira Hospital
Locations (1):
- Faculty of Medicine ,Vajira hospital,Navamindradhiraj University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share in protocol.io

REFERENCES:
- See also: 5. Centers for Disease Control and Prevention. Decontamination and reuse of filtering facepiece respirators — https://www.cdc.gov/coronavirus/2019-ncov/hcp/ppe-strategy/decontamination-reuse-respirators.